CLINICAL TRIAL: NCT04836442
Title: An Integrated Personalized Feedback Intervention for Hazardous Drinkers With Subclinical PTSD
Brief Title: PFI Hazardous Drinkers With Subclinical PTSD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Houston (Other)
Responsible Party: Principal Investigator, Michael J. Zvolensky, Ph.D., Hugh Roy and Lillie Cranz Cullen Distinguished University Professor, University of Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY2021001-AP-PFI
Record Dates: First submitted 2021-04-05; First posted 2021-04-08 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Hazardous Drinking; Posttraumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Ethanol

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alcohol-PTSD-PFI (AP-PFI) (Experimental): Hazardous drinkers with at least subclinical PTSD and elevated AS (N=100) recruited from the community will be randomly assigned to receive Alcohol-PTSD-PFI (AP-PFI) or an active comparison control condition (C-PFI).
  Interventions: Other: Alcohol-PTSD-PFI (AP-PFI)
- Active Comparison Condition (C-PFI) (Other): Participants in the time-matched comparison condition will receive personalized feedback on alcohol use but will not receive PTSD or AS-related personalized feedback. C-PFI will include alcohol-focused components identical to those provided in AP-PFI (e.g., alcohol profiles, normative feedback). Therefore, it will be possible to isolate the impact of personalized PTSD and AS feedback versus personalized alcohol feedback.
  Interventions: Other: Active Comparison Condition (C-PFI)

INTERVENTIONS:
Other: Alcohol-PTSD-PFI (AP-PFI) — Integrated computer-based personalized feedback intervention to specifically target anxiety sensitivity in the context of hazardous drinking and PTSD symptoms. The AP-PFI will focus on feedback about alcohol behavior in the context of PTSD symptoms, AS, and coping-oriented alcohol use.
  Arms: Alcohol-PTSD-PFI (AP-PFI)
Other: Active Comparison Condition (C-PFI) — Participants in the time-matched comparison condition will receive personalized feedback on alcohol use but will not receive PTSD or AS-related personalized feedback. C-PFI will include alcohol-focused components identical to those provided in AP-PFI (e.g., alcohol profiles, normative feedback). Therefore, it will be possible to isolate the impact of personalized PTSD and AS feedback versus personalized alcohol feedback.
  Arms: Active Comparison Condition (C-PFI)

SUMMARY:
The objective of the present study is to assist on a randomized controlled trial (RCT), aimed at developing and testing the efficacy of a novel computer based PFI among hazardous drinkers with at least subclinical posttraumatic stress disorder (PTSD) (i.e., endorsing at least two symptoms in each PTSD symptom cluster) and elevated anxiety sensitivity (AS). The objective of this trial is to examine the feasibility, acceptability, and efficacy of this novel PFI on (1) primary outcomes including drinking motivational factors and alcohol-related behaviors and (2) secondary outcomes including changes in AS and PTSD, and (3) exploring theoretically relevant mediators/moderators. Follow-up assessments will occur at post-test, one-week, and one-month post-intervention. Hazardous drinkers with at least subclinical PTSD and elevated AS (N=100) recruited from the community will be randomly assigned to receive Alcohol-PTSD-PFI (AP-PFI) or an active comparison condition (C-PFI).

DETAILED DESCRIPTION:
Hazardous drinking (i.e., a pattern of alcohol use that increases risk for adverse health consequences) and posttraumatic stress disorder (PTSD) are highly prevalent and commonly co-occurring conditions that are associated with greater disability, mortality, and poor health outcomes as compared to either condition alone. More than 25% of U.S. adults endorse hazardous drinking, which is one of the leading causes of preventable death in the U.S. and globally. Among individuals who engage in hazardous drinking, the prevalence of PTSD is 27% (reflecting 5.81 million people) and individuals who experience PTSD symptoms are roughly three times more likely to endorse hazardous drinking compared to those without PTSD symptomatology. Hazardous drinking-PTSD comorbidity evince bidirectional and transactional effects between PTSD and the maintenance and/or exacerbation of alcohol use. Yet, no empirically supported "gold standard" treatments are available and the most promising interventions are marked by substantive attrition and small effect sizes. Therefore, it is important to consider malleable factors that underlie hazardous drinking-PTSD relations to inform personalized evidence-based interventions among this underserved population.

A transdiagnostic factor for hazardous drinking and PTSD is anxiety sensitivity (AS). AS, defined as the fear of anxiety-related sensations and cognitions, has been positively related to hazardous drinking and coping-oriented drinking motives. Elevated AS has also been implicated in the development and maintenance of PTSD. AS may underlie (i.e., help explain) hazardous drinking-PTSD comorbidity by amplifying PTSD symptomatology and motivating drinking to down regulate such affect. Despite the efficacy of AS interventions for reducing hazardous drinking and PTSD symptoms, an integrated intervention to specifically target AS in the context of hazardous drinking and PTSD symptoms has not been developed or tested. Personalized feedback interventions (PFI) may help to address this gap as they have demonstrated efficacy in reducing hazardous drinking and alcohol-related consequences across various populations. PFI's target misperceptions regarding an individual's behaviors and actual normative behaviors, highlight consequences of these behaviors, and offer strategies for modifying them. Thus, PFIs are brief, cost-effective, easily disseminable, and clinically relevant given low treatment-seeking rates found among hazardous drinkers with PTSD.

Concordant with NIAAA's 2017-2021 Strategic Plan, the objective of the present study is to assist on a randomized controlled trial (RCT) aimed at developing and testing the efficacy of a novel computer based PFI among hazardous drinkers with at least subclinical PTSD (i.e., endorsing at least two symptoms in each PTSD symptom cluster) and elevated AS. The objective of this proposal is to examine the feasibility, acceptability, and efficacy of this novel PFI on (1) primary outcomes including drinking motivational factors and alcohol-related behaviors and (2) secondary outcomes including changes in AS and PTSD, and (3) exploring theoretically relevant mediators/moderators. Follow-up assessments will occur at post-test, one-week, and one-month post-intervention. Hazardous drinkers with at least subclinical PTSD and elevated AS (N=100) recruited from the community will be randomly assigned to receive Alcohol-PTSD-PFI (AP-PFI) or an active comparison condition (C-PFI).

The AP-PFI will focus on feedback about alcohol behavior in the context of PTSD symptoms, AS, and coping-oriented alcohol use, to address the following aims:

Aim 1. Assist on evaluating the feasibility and acceptability of AP-PFI vs. C-PFI.

Evaluate initial metrics of feasibility and efficacy focused on the following:

1. Recruitment/retention rates throughout the duration of the study.
2. Treatment acceptability at post-test, treatment utilization at one-week and one-month follow-up.
3. Initial efficacy at post-test, one-week, and one-month follow-up.

Aim 2. Assist on conducting a RCT to examine the efficacy of AP-PFI vs. C-PFI.

At post-test, participants randomized to AP-PFI (vs. C-PFI) will report:

H1A: Greater motivation/intention to reduce (i.e., from hazardous to non-hazardous) drinking.

H1B: Lower levels of AS.

At one-week and one-month follow-up, participants randomized to AP-PFI (vs. C-PFI) will evince:

H2A: Greater change in rates from hazardous to non-hazardous drinking. H2B: Lower frequency and quantity of alcohol consumption and reduced negative consequences of drinking.

H2C: Lower PTSD symptom severity.

Exploratory Aim 3. Explore mediators and moderators. H3: Effects of AP-PFI (vs. C-PFI) on follow-up outcomes (H2A; H2B; H2C) will be mediated by: (1) motivation/intention to reduce drinking (H1A) and (2) lower levels of AS (H1B).

H4: The effects of AP-PFI (vs. C-PFI) on post-test and one-week and one-month follow-up outcomes will be larger among female (relative to male) participants.

H5: Associations between PTSD and alcohol-related outcomes (e.g., urges, cravings, motivation to reduce drinking, hazardous drinking levels) will be moderated by family history of AUD.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 21 years of age
* Current hazardous drinking pattern (AUDIT scores ≥ 8 for males and ≥ 7 for females; this approach does not exclude persons with alcohol use disorder)
* Lifetime exposure to a DSM-5 Criterion A traumatic event and endorsing at least two symptoms in each DSM-5 PTSD symptom cluster.
* Elevated AS score (1 SD above normative mean)
* Fluent in English

Exclusion Criteria:

* Concurrent alcohol or other substance use treatment
* Current/past bipolar or psychotic disorder
* Current imminent risk of suicidality (i.e., past month ideation with intent or plan)
* Current stable use of prescription opioids/ benzodiazepines/positive urine drug screen
* Current pregnancy
* Inability to provide verbal or written consent
* Breath analysis (Alco-Sensor FST) estimating blood alcohol concentration (BAC) above 0

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-07 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Changes in anxiety sensitivity levels: Short Scale Anxiety Sensitivity Index (SSASI) | administered at one-week and one-month follow-ups
  The Short Scale Anxiety Sensitivity Index utilizes a 5-item Likert scale to measure anxiety sensitivity. The minimum value is "very little" and the maximum value is "Very much". Higher score indicate higher levels of anxiety sensitivity. This index will be used to assess changes in levels of anxiety sensitivity throughout the study. Hypothesis 1b: At post-test, participants randomized to AP-PFI (vs. C-PFI) will report lower levels of anxiety sensitivity.
Changes in motivation/intention to reduce drinking: The Alcohol Ladder | administered at one-week and one-month follow-ups
  The Alcohol Ladder is a one-item, reliable measure that assesses an individual's motivation to change their alcohol use. The ladder includes 10 rungs and asks participants to rate readiness to change their drinking habits by asking "Each rung of this ladder shows where a person might be in thinking about changing their drinking. Select the number that best matches where you are now.". The higher participants rate themselves on the ladder, the higher their readiness to change their drinking. This measure will be used to assess changes in motivation to reduce drinking throughout the study. Hypothesis 1a: At post-test, participants randomized to AP-PFI (vs. C-PFI) will report greater motivation/intention to reduce (i.e., from hazardous to non-hazardous) drinking.
Changes in hazardous drinking patterns: Alcohol Use Disorders Identification Test | administered at baseline, one-week and one-month follow-ups
  The alcohol use disorder identification test assesses drinking patterns and related consequences, and is valid, reliable, and demonstrates excellent sensitivity to detect potentially hazardous drinkers. Although all participants will be screened with the full measure, the first three items will be administered at follow-ups to evaluate hazardous alcohol use over time. Hypothesis 2a: At one-week and one-month follow-up, participants randomized to AP-PFI (vs. C-PFI) will evince greater change in rates from hazardous to non-hazardous drinking.
Changes in frequency and quantity of alcohol consumption: Timeline Follow-Back | administered at baseline, one-week and one-month follow-ups
  The Timeline Follow-Back (TLFB) is a calendar-based questionnaire that collects information regarding alcohol consumption over the past 30 days and is a reliable measure. It will be used to assess the changes in frequency and quantity of alcohol consumption throughout the study. Hypothesis 2b: at one-week and one-month follow-up, participants randomized to AP-PFI (vs. C-PFI) will evince lower frequency and quantity of alcohol consumption and reduced negative consequences of drinking.
Changes in PTSD symptom severity: The Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5) | administered at baseline, one-week and one-month follow-ups
  The Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5) measures PTSD symptom severity as it relates to the "worst" traumatic event endorsed throughout the participant's lifespan. The PCL-5 is a 20-item self-report measure that assesses the 20 DSM-5 symptoms of PTSD. A total symptom severity score (range - 0-80) can be obtained by summing the scores for each of the 20 items, whereas higher scores represent higher symptom severity. It will be administered to participant throughout the study in order to assess changes in posttraumatic stress disorder symptom severity. Hypothesis 2c: At one-week and one-month follow-up, participants randomized to AP-PFI (vs. C-PFI) will evince lower PTSD symptom severity

SECONDARY OUTCOMES:
Evaluate the feasibility and acceptability of AP-PFI vs. C-PFI: Treatment Credibility/Expectancy Questionnaire | administered at one-month follow-up
  The acceptability of the intervention (i.e., AP-PFI) will be assessed via the Treatment Credibility/Expectancy Questionnaire (TCEQ). This measure is a reliable index that will be used to assess perceptions of treatment credibility/expectancies about treatment, including satisfaction, acceptability of AP-PFI relative to control. Additionally, it will assess how participants think the intervention will be successful in terms of reducing alcohol use, PTSD symptoms, and anxiety sensitivity, while also assessing anticipated reductions in alcohol use, PTSD symptoms, and anxiety sensitivity (0-100%).
Evaluate the moderating role of family history of AUD on PTSD and alcohol-related outcomes | Administered at baseline
  Will be assessed via the Alcohol History Measure (AHM), a 11-item questionnaire that collects information on a participant's history of alcohol use, including familial history, consequences associated with use, and age of first use.

CONTACTS AND LOCATIONS:
Locations (1):
- Anxiety and Health Research Lab- Substance Use Treatment Clinic, Houston, Texas, United States